CLINICAL TRIAL: NCT03062501
Title: Protocol for the Administration of Hydroxyurea During Painful Vaso-occlusive Crisis in Sickle Cell Anemia
Brief Title: Hydroxyurea in the Emergency Room to Lessen Pain in Sickle Cell Crisis
Acronym: HELPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Estadual de Hematologia Arthur de Siqueira Cavalcanti (Other)
Responsible Party: Principal Investigator, CLARISSE LOBO, PI, Instituto Estadual de Hematologia Arthur de Siqueira Cavalcanti
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hemorio 397/16
Record Dates: First submitted 2017-01-30; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Anemia, Sickle Cell; Anemia; Sickle-Cell, With Crisis
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Hydroxyurea) (No Intervention): Patients in VOC will be treated according to the center's usual practice and analgesia protocol.
- Hydroxyurea (Experimental): Patients in VOC will receive up to three daily doses of 30-40 mg / kg hydroxyurea.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Patients hospitalized for uncomplicated pain crisis with a pain scale of ≥ 6 during the last 24 hours will receive a dose of 30-40 mg / kg hydroxyurea. This same dose of hydroxyurea will be repeated at 24 h and 48 h after the first dose of hydroxyurea, with dose suspension if the patient is discharged within 48 hours. Patients will also receive the center's usual practice and analgesia protocol.
  Arms: Hydroxyurea

SUMMARY:
This study will investigate the safety, tolerability and potential for the use of up to three daily doses of 30-40 mg/kg HU (daily) upon hospitalization for painful vaso-occlusive crises .

DETAILED DESCRIPTION:
Sickle cell anemia (SCA) is a hereditary hemoglobinopathy; complications of the disease include, spleen enlargement, acute chest syndrome, pulmonary hypertension, stroke and cumulative damage to multiple organs, and painful vaso-occlusive crises (VOC). In Brazil, about 3,500 children are born each year with DF, and the number of individuals with sickle cell disease (DF) in the country is estimated between 25,000 and 30,000 (ANVISA 2012; BRAZIL, 2012).

Hydroxyurea (HU, or hydroxycarbamide) is the only drug approved to date by the American FDA for use in adults with sickle cell disease. The drug modifies the disease process, improving hematological parameters and the hospitalization time of patients, as well as the frequency of vaso-occlusive crises.In addition to its proven effects during chronic use, experimental data indicate that HU has immediate anti-inflammatory effects.

In addition to its proven effects during chronic use, experimental data indicate that HU has immediate anti-inflammatory effects. This study will investigate the safety, tolerability and potential for the use of up to three daily doses of 30-40 mg/kg HU (daily) upon hospitalization for VOC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of homozygous sickle cell anemia (HbSS).
* Hospitalization due to onset of uncomplicated vaso-occlusive crisis (with pain scale≥6 within the last 24 h), confirmed by clinical evaluation.
* Documented and written informed consent

Exclusion Criteria:

* Confirmed or suspected pregnancy.
* Initiation of painful crisis> 72h.
* Blood transfusion during the last 8 weeks.
* Admission to Emergency Room due to pain in the last 4 weeks.
* Neutrophil count <2.5 x 109/L or platelet count <95.0 x 109 / L or Hb <4.5 g / dL
* Weight <38 Kg or> 95 Kg.
* Interval longer than 8h since arrival at center.
* Non-consent to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | up to 15 days post last dose
  as assessed by CTCAE version 4.03
Number of participants with altered laboratory values related to treatment | up to 15 days post last dose

SECONDARY OUTCOMES:
Time until hospital discharge | Average, up to 7 days post admission
Total opioid use (mg of IV morphine) | From study inclusion until hospital discharge (average, up to 7 days post admission)
Pain score | From admission until hospital discharge (average, up to 7 days post admission)
  Numeric pain score rating (0 to 10; 0 = no pain, 10 = worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Hemorio, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No